CLINICAL TRIAL: NCT01310153
Title: Effect of Supine or Prone Position at Delivery on Respiratory Outcomes in Full-Term Infants Following Elective Caesarean Birth
Brief Title: Effect of Supine or Prone Position After Caesarean Birth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Orna Rosen, Asst Prof., Dept of Pediatrics (Neonatology), Montefiore Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 06-09-409
Record Dates: First submitted 2011-03-04; First posted 2011-03-08 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Respiratory Distress; Transient Tachypnea of the Newborn; Delayed Transition of the Newborn; Persistent Pulmonary Hypertension
MeSH Terms: conditions — Dyspnea; Transient Tachypnea of the Newborn | interventions — Prone Position; Supine Position

ARMS (2):
- Prone Positioning (Active Comparator): Newly born infant placed in prone position (face up) for the first 30 60 seconds of life after delivery by Cesarean birth.
  Interventions: Procedure: prone positioning
- Supine Positioning (Active Comparator): newly born infant placed in supine position (face down) for the first 30 60 seconds of life after delivery by Cesarean birth.
  Interventions: Procedure: Supine

INTERVENTIONS:
Procedure: prone positioning — newborn babies in prone positioning
  Arms: Prone Positioning
Procedure: Supine — newborn babies in supine positioning
  Arms: Supine Positioning

SUMMARY:
Respiratory Distress is a frequent clinical diagnosis of babies delivered by elective Caesarean birth. There has been no study comparing the efficacy of immediately positioning a newly born infant prone vs. supine for the first 30 60 seconds of life after delivery by Caesarean birth.

DETAILED DESCRIPTION:
This study hypothesizes that when the infant is prone they will have postural drainage, better dorsal lung expansion, less vagal response from suctioning and less agitation secondary to the righting reflex.

This study will compare 1033 term babies divided by randomization into two groups prone and supine. During the study, care givers will monitor and record incidence and severity of Respiratory Distress, Use of FiO2 or respiratory support, admissions to NICU.

ELIGIBILITY:
Inclusion Criteria:

* Any woman not in labor who are undergoing elective Cesarean birth at term, 37 to 41 completed weeks gestation.

Exclusion Criteria:

* any woman with prior rupture of membranes
* diabetes mellitus, gestational diabetes,
* any woman receiving sedation
* using medication such as Demerol, magnesium sulfate or general anesthesia
* any woman who has a known drug history
* any known macrosomia
* known congenital anomalies or meconium stained fluid
* any woman with illnesses such as maternal fever, chorioamnionitis, severe neonatal distress
* any woman with compromised infant at delivery
* oligohydramnios
* history of antenatal steroids.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2006-09; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Orna Rosen, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Jack D. Weiler Hospital of the Albert Einstein College of Medicine, The Bronx, New York, United States